CLINICAL TRIAL: NCT05429125
Title: A Randomized Comparison Between the Flexible Tip Bougie vs Tube With Stylet for First-attempt Intubation Success With the C-MAC Videolaryngoscopy in Patients With Anticipated Difficult Airway
Brief Title: Flexible Tip Bougie vs Tube With Stylet for Intubation With Videolaryngoscopy.
Acronym: VIFLEXTIPOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Professor, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIDEOLAR-FLEXTIP-OR
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Intubation; Difficult or Failed
Keywords: intubation; difficult airway; videolaryngoscope; operating room; Awake intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal Tube with Stylet (Active Comparator): Patients randomised to Endotracheal Tube with Stylet will be intubated with a Videolaryngoscopy and with an endotracheal tube + stylet.
  Interventions: Device: Endotracheal Tube with Stylet
- Flexible Tip Bougie (Active Comparator): Patients randomised to Flexible Tip Bougie will be intubated with a Videolaryngoscopy and with a Flexible Tip Bougie.
  Interventions: Device: Flexible Tip Bougie

INTERVENTIONS:
Device: Endotracheal Tube with Stylet — Patients randomised to Endotracheal Tube with Stylet will be intubated with a Videolaryngoscopy and with an endotracheal tube + stylet.
  Arms: Endotracheal Tube with Stylet
Device: Flexible Tip Bougie — Patients randomised to Flexible Tip Bougie will be intubated with a Videolaryngoscopy and with a Flexible Tip Bougie.
  Arms: Flexible Tip Bougie

SUMMARY:
Although VLs improve glottic visualization, on many occasions it may not be accompanied by intubation at the first attempt, because the endotracheal tube has to pass a sharp angle to enter the trachea. To avoid this limitation, a new flexible tip bougie is designed to flexibly navigate the distal tip and help facilitate precise insertion of the endotracheal tube in the trachea. The flexible tip bougie has an integrated slider along the surface which moves the tip anterior and posterior while the pre-curved distal portion of shaft allows the angulation to provide anterior flexion. This new flexible tip bougie could be used as a rescue when first intubation failure using the videolaryngoscopy, or as a first option to improve the percentage of patients intubated at the first attempt.

DETAILED DESCRIPTION:
The purpose of this prospective randomized study is to compare successful intubation on the first attempt with the new flexible tip bougie versus endotracheal tube with stylet during awake intubation with videolaryngoscopy in patients with anticipated difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients with anticipated difficult airway requiring intubation under with a videolaryngoscopy
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Pregnancy
* age <18 years
* refusal of the patient
* patient's respiratory failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the first attempt intubation success rate (percentage) | During intubation
  To compare the difference in the first attempt intubation success rate (percentage) with the two differents devices compared.

SECONDARY OUTCOMES:
Difference in the overall intubation success rate (percentage) | During intubation
  To compare the difference overall intubation success rate (percentage) with the two differents devices compared.
Difference in the incidence of complications (percentage) | Participants will be followed from the beginning of the intervention to 30 minutes after the intervention
  To compare the difference in complications (percentage) with the two different devices compared:
  Hypoxemia (SpO2) < 90 %, Hypoxemia severe (SpO2) < 80 %, Hypotension defined as systolic blood pressure less than 80 mm Hg, Severe hypotension defined as systolic blood pressure less than 65 mm Hg, Cardiac arrest, death during intubation, Moderate or difficult intubation, oesophageal intubation, pulmonary aspiration, dental injuries.
Difficulty of intubation | During intubation
  Operator-assessed subjective difficulty of intubation by means of a special analogue numerical scale from 0 to 10, where 0=no subjective difficulty and 10=maximal subjective difficulty
Modified Cormack-Lehane grade of glottic view | During intubation
  Modified Cormack-Lehane grade of glottic view:
  I: full view of the glottis IIa: partial view of the glottis IIb: arytenoid or posterior part of the vocal cords just visible III: only epiglottis visible IV: neither glottis nor epiglottis visible
Additional airway equipment | During intubation
  Need for additional airway equipment
Number of intubation attempts | During intubation
  Number of intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada Muñiz, Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved T ypes of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Ruetzler K, Smereka J, Abelairas-Gomez C, Frass M, Dabrowski M, Bialka S, Misiolek H, Plusa T, Robak O, Aniolek O, Ladny JR, Gorczyca D, Ahuja S, Szarpak L. Comparison of the new flexible tip bougie catheter and standard bougie stylet for tracheal intubation by anesthesiologists in different difficult airway scenarios: a randomized crossover trial. BMC Anesthesiol. 2020 Apr 20;20(1):90. doi: 10.1186/s12871-020-01009-7. PMID 32312225
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096